CLINICAL TRIAL: NCT07261397
Title: The Effect of the Nurse-Led ROOTS Program and Soft Skills Training on Emotional Regulation to Prevent Bullying in High School Students in Bandung City: A Quasi-Experimental
Brief Title: Nurse-Led ROOTS-Soft Skills Intervention for Bullying Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NURS-202511.01
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Bullying Behavior; Emotional Regulation Difficulties; Adolescent Mental Health
Keywords: Bullying Prevention; Emotional Regulation; Empathy; High School Students; Nurse-Led Intervention
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Students are assigned to either the intervention group receiving the ROOTS and Soft Skills sessions or a control group receiving school-as-usual activities. The intervention lasts 8 weeks with pre- and post-assessments.
Who Masked: Outcomes Assessor
Masking Description: Participants and school staff are aware of group allocation, but outcome assessors are blinded to minimize measurement bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants receive the Nurse-Led ROOTS Program combined with Soft Skills Training. This eight-week program, facilitated by the school nurse and a teacher, includes peer-led leadership activities, emotion regulation exercises, assertive communication, cognitive reappraisal, and empathy training to prevent bullying and improve emotional regulation.
  Interventions: Behavioral: Nurse-Led ROOTS Program and Soft Skills Training
- Control Group (No Intervention): Participants in this arm will receive standard care provided at the school without additional psychological intervention.

INTERVENTIONS:
Behavioral: Nurse-Led ROOTS Program and Soft Skills Training — A structured, eight-week program delivered once per week (60-90 minutes/session) by the school nurse and supported by teachers. Core components include:
  Program orientation and group norms
  Peer leadership and assertive communication
  Emotional awareness and labeling
  Expression management and self-control
  Cognitive reappraisal exercises
  Empathy and perspective-taking
  Peer-led positive values campaign
  Reflection, feedback, and skill consolidation
  Arms: Intervention Group

SUMMARY:
This study aims to evaluate the effect of a nurse-led intervention combining the ROOTS program and soft skills training on emotional regulation and bullying prevention among high school students in Bandung, Indonesia. Bullying remains a major concern in schools and is closely linked to emotional difficulties, poor coping skills, and limited empathy. Strengthening students' emotional regulation is an evidence-based strategy to reduce aggressive behaviors and promote safer school environments.

In this study, trained school nurses will deliver an integrated intervention consisting of sessions on identifying emotions, managing stress, developing empathy, communicating effectively, and resolving conflicts. The program is designed to help students better understand their emotions, control impulsive reactions, and build positive relationships with peers. These skills are expected to reduce the risk of bullying-both as perpetrators and as victims.

The research uses a quasi-experimental design involving two high schools in Bandung. One school will receive the nurse-led intervention, while the comparison school will continue routine school activities. Students who meet inclusion criteria and provide consent/assent will participate in pre- and post-intervention assessments. The primary outcome is improvement in emotional regulation scores. Secondary outcomes include bullying behavior, empathy, and student perceptions of the school climate.

All activities will follow ethical guidelines, including confidentiality, voluntary participation, and the right to withdraw at any time. The study seeks to provide evidence on how nurses can contribute to mental health promotion in schools and support sustainable, school-based bullying prevention strategies.

DETAILED DESCRIPTION:
This study investigates a structured, nurse-led intervention that integrates the ROOTS program with soft skills training to enhance emotional regulation as a strategy to prevent bullying among adolescents. The intervention consists of multiple structured sessions delivered over several weeks, focusing on emotional awareness, stress management, empathy development, communication strategies, and problem-solving skills. The program was adapted for Indonesian high school students and aligned with the role of school nurses in mental health promotion.

A quasi-experimental non-randomized design will be used. Two high schools in Bandung will participate: one serving as the intervention site and the other as the comparison site. Participants will be students in grades 10-11 who consent to join the study. Pre-intervention assessments will measure emotional regulation (primary outcome) and bullying behaviors, empathy, and school climate (secondary outcomes). After the intervention sessions are completed, the same measures will be reassessed.

The study aims to generate evidence on the feasibility and effectiveness of a nurse-led emotional and social skills program delivered in school settings. Findings are expected to inform future mental health strategies, support the integration of nurses into school-based preventive services, and contribute practical recommendations for bullying prevention policies.

ELIGIBILITY:
Inclusion Criteria

* Adolescents aged 14-18 years
* Enrolled in participating secondary schools
* Willing to provide assent, with parental/guardian consent
* Able to understand and communicate in the local language (e.g., Indonesian or English)
* Identified as having mild to moderate difficulties in emotional regulation or at risk for anxiety/depression based on school screening Exclusion Criteria
* Severe psychiatric conditions requiring immediate clinical intervention (e.g., psychosis, severe depression with suicidal intent)
* Currently receiving structured psychological or psychiatric treatment for emotional regulation or mental health conditions
* Cognitive or developmental disabilities that would prevent meaningful participation in group activities
* Non-consent from parent/guardian or the participant

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-05 (Actual)

PRIMARY OUTCOMES:
Emotional Regulation | Pre-intervention (week 0) and post-intervention (week 8)
  Emotional regulation ability is measured using the Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA), a 10-item instrument rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 10 to 50, with higher total scores indicating better overall emotional regulation ability. Changes in the total ERQ-CA score from pre-intervention (week 0) to post-intervention (week 8) are used to evaluate the extent to which the intervention improves participants' capacity to manage and express their emotions adaptively.

CONTACTS AND LOCATIONS:
Overall Officials: Iyus Yosep, Principal Investigator — Universitas Padjadjaran
Locations (1):
- SMA Al Marwah and MAN Kota Bandung, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The dataset contains sensitive mental health information from adolescents, and institutional policies prohibit the release of such de-identified data to external researchers.